CLINICAL TRIAL: NCT03409536
Title: Evaluation of the Diagnostic Threshold of SSEP of Brachial Plexus Injury
Brief Title: Somatosensory Evoked Potential (SSEP) Monitoring for Brachial Plexus Injury
Status: Completed | Type: Observational
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Principal Investigator, Jason Chui, Assistant Professor, Anesthesiologist, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Other Study IDs: SSEP BPI
Record Dates: First submitted 2018-01-18; First posted 2018-01-24 (Actual); Last update posted 2020-02-19 (Actual); Status verified 2020-02

CONDITIONS: Brachial Plexus Injury; Peripheral Nerve Injuries
Keywords: SSEP Monitoring; Diagnostic threshold
MeSH Terms: conditions — Peripheral Nerve Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- SSEP Monitoring: participants will receive a brachial plexus block for their surgery and will be monitored for brachial plexus injury using the automated SSEP monitor.
  Interventions: Device: SSEP monitoring

INTERVENTIONS:
Device: SSEP monitoring — Participants will be monitored using the SSEP device both before and after induction of a brachial plexus block.

SUMMARY:
Brachial plexus block is a common regional anesthesia technique which is performed by anesthesiologists to anesthetize the arm for surgery. In this study, we are investigating the relationship between the nerve conduction (induced by brachial plexus block) and the patients' symptoms before and after the brachial plexus block. We will attach a nerve conduction device (SSEP device) to monitor the patients' arm conduction and we will assess the patients' symptoms simultaneously.

DETAILED DESCRIPTION:
Perioperative peripheral nerve injury (PNI) is an under-recognized and under-investigated complication of general anesthesia and continues to impact postoperative recovery resulting in patient disability malpractice claims.(1-5) In the American Society of Anesthesiologists (ASA) Closed Claims Analysis (published in 1999), PNI was the second most common cause of claims other than death. (6-7) This claim pattern has remained essentially unchanged over the past 3 decades and the average settlement was $123,000 US Dollar/claim (unpublished data from ASA closed claims analysis). The overall incidence of PNI varies across different surgical procedures, and it is significantly affected by the underlying patient comorbidities and pre-existing peripheral neuropathy. Despite considerable implications of PNI to both the patients and clinicians, little progress has been made in the past three decades in developing a reliable intraoperative monitoring technique for its early detection and prevention. SSEP monitoring has long been used in neurology as a means to diagnose peripheral neuropathy and has been used for the early detection of intraoperative PNI caused by improper patient positioning. A few retrospective studies have found that reversal of intraoperative SSEP signal changes (e.g. correct the patient's arm position in the event of a positioning related peripheral nerve compromise) prevented postoperative neuropathy, suggesting SSEP could be used to detect intraoperative PNI and that prompt intervention could reverse neurological injury (8-10). However, to date, there has not been a study that clearly defines how the magnitudes of SSEP changes relate to the severity of peripheral nerve dysfunction. Due to this lack of information, the current thresholds that are used for diagnosing PNI in a variety of surgical procedures are largely based on the results of SSEP monitoring in spinal cord injury. The traditional diagnostic criteria (used in spinal cord injury) might not be applicable for PNI. Fundamentally, there is also a lack of a clinical study that defines significant and non-significant changes for PNI. Most current available evidence regarding SSEP in PNI is retrospective and mainly derived from patients being monitored for spinal cord or cerebral injury during neurosurgical procedures. The lack of well-validated diagnostic criteria is one of the key issues in preventing the use of SSEP for monitoring peripheral nerves during surgery. As such, further studies are required to characterize the relationship between SSEP changes and peripheral nerve dysfunction and re-define the threshold (or cut-off values) for significant SSEP change for PNI.

This is a prospective cohort study to evaluate the relationship between the peripheral nerve dysfunction, and SSEP signal changes in patients who will receive a brachial plexus block for their surgical procedure. Brachial plexus block is a regional anesthesia technique routinely performed by anesthesiologists where the nerves in the arm are blocked with local anesthetics to prohibit movement and sensation. In LHSC, the average brachial plexus block performed is around 10-15 patients/day for various upper limb surgeries. In this study, the patients with brachial plexus block will be used as a model of brachial plexus injury to assess the relationship between intraoperative brachial plexus injury and the SSEP changes. Brachial plexus block in awake patients is an attractive model to study brachial plexus injury, because it provides transient and progressive de-afferentation state of brachial plexus dysfunction (mimicking brachial plexus injury), allows for real-time assessment of the relationship between clinical symptoms and SSEP changes (awake patients), and overcomes obvious practical limitations of investigating intraoperative PNI (small sample size of patients with intraoperative brachial plexus injury). In this study, 50 consecutive patients who required a brachial plexus block for their surgery, will be recruited. This study will be performed in the "Block Room" of either London Health Science Centre or St Joesph Hospital, London, Ontario. After obtaining informed consent, an independent assessor (hand specialist) will perform a baseline assessment of the sensory and motor function of the upper limb. The sensory function will be quantified by a two-point discrimination test in each dermatome. The motor function will be quantified by the motor score in each myotome. The patients will be attached to the automated SSEP monitor to obtain baseline upper limb SSEP signals. Median, ulnar and radial nerves will be monitored. After satisfactory baseline SSEP recordings have been obtained, a brachial plexus block will be performed in the usual fashion to achieve complete sensory and motor blockage (approx. 30 min). This provides a unique experimental condition to assess the relationship between the brachial plexus dysfunction and the SSEP signal changes. An independent assessor (hand specialist) will re-assess the patients' sensory and motor function every 5 minutes (up to 30 minutes during the onset of the block). SSEP recording will be concomitantly obtained. A total of 300 data pairs (6 data pairs for each patient) will be obtained for analysis. In this study, the Evoked Potential Assessment Device (EPAD®, SafeOp Surgical, Hunt Valley, MD) SSEP machine will be used. It is a novel, simplified, automated SSEP monitoring device (FDA approved), designed to detect intraoperative PNI. The key features of EPAD® are that only the surface adhesive electrodes (i.e. no subdermal needle electrodes) will be used, as well as there is newly artifact rejection and optimization algorithm that permit SSEP recording in awake patients.

Prior to performing the brachial plexus block in the "Block room", a complete neurological examination will be performed including motor score and 2-point discrimination test. Eligible patients will be recruited after obtained informed consent. The baseline SSEP of the participants will be recorded using the EPAD@ device. After the participants received the brachial plexus block (as part of their standard of care), the participants will be monitoring the progressive changes of SSEP signals while the effect of brachial plexus block gradually onset (usually takes around 30 minutes). An independent assessor (hand specialist blinded to the SSEP results) will concomitantly re-assess the patients' sensory and motor function every 5 minutes (up to 30 minutes during the onset of the block).

The primary analysis will be on describing the relationship between the severity of the neurological deficits (impaired sensory and/or motor function) and SSEP changes (amplitude and/or latency changes). Secondarily, an optimal cut-off limit using Youden index and/or logistic regression-derived likelihood ratio functions will be determined. A Receiver-operating-curve for the new cut-off limits will be assessed. REDCapTM will be used for electronic data collection and STATA (version 14) will be used for statistical analysis in all the studies. These new cut-off limits in comparison with conventional criteria in our subsequent clinical studies will be compared.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients who are scheduled to have elective upper limb surgeries and require a brachial plexus block as part of their standard of care.

Exclusion Criteria:

* Patients unable to perform a complete neurological examination (e.g. dementia, upper limb fracture).
* Patients who refuse to participate or unable to provide informed consent.
* Patients who are contraindicated for SSEP monitoring.
* Patients who have known pre-existing peripheral neuropathy or brachial plexus injury.
* Patients who are contraindicated to brachial plexus block.
* Patients who are not undergoing brachial plexus block for their procedures (e.g. elective C5 nerve root block).
* Patients who had failed brachial plexus block.

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patients who are scheduled to have elective upper limb surgeries and require a brachial plexus block as part of their standard of care.
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Neurological symptoms (including sensory and motor) | 0-30 minutes after receiving the brachial plexus block
  Neurological symptoms (including sensory and motor)

CONTACTS AND LOCATIONS:
Overall Officials: Jason Chui, MBChB, Principal Investigator — London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Locations (1):
- St Joeshp Hospital, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wojtkiewicz DM, Saunders J, Domeshek L, Novak CB, Kaskutas V, Mackinnon SE. Social impact of peripheral nerve injuries. Hand (N Y). 2015 Jun;10(2):161-7. doi: 10.1007/s11552-014-9692-0. PMID 26034424
- [Background] Grocott HP, Clark JA, Homi HM, Sharma A. "Other" neurologic complications after cardiac surgery. Semin Cardiothorac Vasc Anesth. 2004 Sep;8(3):213-26. doi: 10.1177/108925320400800304. PMID 15375481
- [Background] Sharma AD, Parmley CL, Sreeram G, Grocott HP. Peripheral nerve injuries during cardiac surgery: risk factors, diagnosis, prognosis, and prevention. Anesth Analg. 2000 Dec;91(6):1358-69. doi: 10.1097/00000539-200012000-00010. No abstract available. PMID 11093980
- [Background] Tajiri O, Tateda T, Sugihara H, Yokoyama H, Nishikido O, Mukumoto C. [Brachial plexus neuropathy following open-heart surgery]. Masui. 2004 Apr;53(4):407-10. Japanese. PMID 15160668
- [Background] Fitzgerald M, McKelvey R. Nerve injury and neuropathic pain - A question of age. Exp Neurol. 2016 Jan;275 Pt 2:296-302. doi: 10.1016/j.expneurol.2015.07.013. Epub 2015 Jul 26. PMID 26220898
- [Background] Kroll DA, Caplan RA, Posner K, Ward RJ, Cheney FW. Nerve injury associated with anesthesia. Anesthesiology. 1990 Aug;73(2):202-7. doi: 10.1097/00000542-199008000-00002. PMID 2382845
- [Background] Cheney FW, Domino KB, Caplan RA, Posner KL. Nerve injury associated with anesthesia: a closed claims analysis. Anesthesiology. 1999 Apr;90(4):1062-9. doi: 10.1097/00000542-199904000-00020. PMID 10201678
- [Background] Larson SJ, Gandhoke GS, Kaur J, et al. Incidence of position related neuropraxia in 4489 consecutive patients undergoing spine surgery. Role of SSEP monitoring? Journal of Neurosurgery 2016; 124 (4): A1182
- [Background] Ying T, Wang X, Sun H, Tang Y, Yuan Y, Li S. Clinical Usefulness of Somatosensory Evoked Potentials for Detection of Peripheral Nerve and Brachial Plexus Injury Secondary to Malpositioning in Microvascular Decompression. J Clin Neurophysiol. 2015 Dec;32(6):512-5. doi: 10.1097/WNP.0000000000000212. PMID 26629760
- [Background] Araus-Galdos E, Delgado P, Villalain C, Martin-Velasco V, Castilla JM, Salazar A. Prevention of brachial plexus injury due to positioning of patient in spinal surgery. Value of multimodal intraoperative neuromonitoring (IONM). Clinical Neurophysiology 2011; 122: S113
- [Derived] Chui J, Freytag A, Glimore G, Dhir S, Rachinsky M, Murkin J. A novel approach of using brachial plexus blockade as an experimental model for diagnosis of intraoperative nerve dysfunction with somatosensory evoked potentials: a blinded proof-of-concept study. Can J Anaesth. 2021 Jul;68(7):1018-1027. doi: 10.1007/s12630-021-01975-7. Epub 2021 Mar 31. PMID 33791897